CLINICAL TRIAL: NCT06691893
Title: A Randomized Controlled Trial to Evaluate the Efficacy of Immobilized Lipase (RELiZORB) During Enteral Nutrition in Patients With Exocrine Pancreatic Insufficiency Secondary to Acute Pancreatitis
Brief Title: Evaluating the Efficacy of RELiZORB in Managing Exocrine Pancreatic Insufficiency in Tube-fed Pancreatitis Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Alcresta Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, Casey M. Luckhurst, Physician, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2024p002758
Record Dates: First submitted 2024-11-13; First posted 2024-11-18 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Exocrine Pancreatic Insufficiency (EPI); Pancreatitis
Keywords: exocrine pancreatic insufficiency; pancreatitis; RELiZORB; lipase; enteral nutrition
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency; Pancreatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- No RELiZORB (No Intervention): Patients will receive tube feeds (via nasogastric or nasojejunal tube) without the use of RELiZORB
- RELiZORB (Experimental): Patients will receive tube feeds (via nasogastric or nasojejunal tube) with the use of RELiZORB
  Interventions: Device: RELiZORB

INTERVENTIONS:
Device: RELiZORB — RELiZORB (immobilized lipase) is a therapeutic device designed to enhance fat absorption in patients receiving enteral tube feedings. It works by hydrolyzing fats found in enteral formulas. RELiZORB is a single-use cartridge that connects in-line with enteral feeding sets. It contains lipase covalently bound to small polymer beads, forming a complex called iLipase, which remains within the cartridge. As the enteral formula passes through the cartridge, its fat content is hydrolyzed upon contact with iLipase. This process is especially beneficial for the absorption of long-chain polyunsaturated fatty acids, which require hydrolysis by pancreatic lipase for proper intestinal absorption. RELiZORB is compatible with a wide variety of commercially available enteral formulas.
  Other Names: Immobilized Lipase
  Arms: RELiZORB

SUMMARY:
This research aims to improve the management of exocrine pancreatic insufficiency (EPI), a condition that can develop after pancreatitis, a painful inflammation of the pancreas. EPI occurs when the pancreas does not produce enough enzymes to help the body properly digest food. While pancreatic enzyme replacement therapy (PERT) is commonly used to manage EPI symptoms, it can be challenging for people who rely on feeding tubes. RELiZORB, could help these patients by simplifying the delivery of the enzymes they need. However, RELiZORB has only been studied in people with EPI caused by cystic fibrosis, so its effectiveness in pancreatitis patients remains unknown. This study aims to determine whether RELiZORB is effective for individuals requiring feeding tube support after pancreatitis.

DETAILED DESCRIPTION:
Acute pancreatitis remains one of the leading gastrointestinal causes of hospital admission in the United States. While most cases of pancreatitis are mild and resolve without further complications, approximately 20% progress to necrotizing pancreatitis, and 10% may develop chronic pancreatitis. Although significant attention has been given to the acute management of necrotizing pancreatitis, there is a growing focus on diagnosing and managing the long-term complications of pancreatitis. Exocrine pancreatic insufficiency (EPI) is a known complication following acute pancreatitis, with even higher rates observed in cases of necrotizing pancreatitis and chronic pancreatitis. Diagnosing and managing EPI is critical, as it has significant implications for patient outcomes and mortality. Despite this, EPI remains underdiagnosed, prompting the publication of multiple guidelines aimed at improving its diagnosis and treatment. The standard treatment for EPI is oral pancreatic enzyme replacement therapy (PERT). While PERT regimens have proven effective, their use in patients requiring tube feeding is often impractical. Immobilized lipase (RELiZORB) offers potential advantages for patients needing enteral nutrition support due to its ease of use, which can improve compliance. Studies have demonstrated that RELiZORB is safe, well-tolerated, and effective at improving fatty acid absorption. However, these studies were conducted in patients with cystic fibrosis (CF). Unlike CF, pancreatitis is an acute disease with dynamic physiological changes. Additionally, the goal for patients with EPI due to pancreatitis is to resume full oral nutrition without relying on enteral feeding. Therefore, further studies are needed to evaluate the efficacy and impact of RELiZORB in this population.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with moderate or severe exocrine pancreatic insufficiency (EPI), as defined using the Pancreatic Exocrine Insufficiency Questionnaire (PEI-Q) symptom score of 1.4 or greater.
* Patient diagnosed with acute, recurrent acute pancreatitis or subacute pancreatitis. Subacute pancreatitis is defined as recent diagnosis of acute pancreatitis with sequelae of the acute episode including infection, pseudocyst, walled-off pancreatic necrosis.
* Patient is currently admitted to the hospital at the time of study enrollment.
* Patient requiring at least 50% of daily caloric and fluid intake through enteral tube feeds.
* Patient is able and willing to provide informed consent.

Exclusion Criteria:

* Patient with chronic pancreatitis
* Patient is currently intubated and unable to provide consent
* Patient with active gastrointestinal tract cancer
* Patient requiring less than 50% of nutritional support at time of enrollment
* Patient is unable to tolerate any form of enteral nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2027-04-15 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
Pancreatic Exocrine Insufficiency Questionnaire (PEI-Q) | Measured at 14 days from randomization
  The PEI-Q is an 18-item Patient-Reported Outcome (PRO) questionnaire designed to help individuals with pancreatic exocrine insufficiency (PEI) assess their symptoms and the impact on their health-related quality of life. Created and validated by Adelphi Values UK in collaboration with Abbott, the PEI-Q is available for use in clinical studies without the need to purchase a license. The scoring system ranges from 0 to 4, with higher scores indicating more severe symptoms. A score between 0.6 and 1.4 reflects mild PEI, 1.4 to 1.8 indicates moderate PEI, and a score of 1.8 or higher signifies severe or poorly controlled PEI.
  Our primary outcome measure is examining the change in baseline PEI-Q symptom score.

SECONDARY OUTCOMES:
Time to treatment failure | Measured up to 14 days from randomization
  Treatment failure is defined as no change from baseline or worsening of the PEI-Q symptom score.
Biochemical Profile | Measured at 30, 60, and 90 days from randomization
  Change in baseline biochemical profile including Omega 3 Index, Fat-Soluble Vitamins (A, D, E, K), Albumin, Pre-albumin, and C-Reactive Protein.
Stool Assessment | Measured at 30, 60, and 90 days from randomization
  Stool consistency and other features indicative of malabsorption (steatorrhea) will be assessed using the Bristol Stool Scale. Patients will also report the presence of steatorrhea (fatty, oily stools) in a stool log.
  The Bristol Stool Scale is a medical tool used to classify and describe the form of human feces. It consists of seven types of stool, each representing a different consistency or appearance. Types 1 and 2 indicate constipation, while types 6 and 7 indicate diarrhea. Types 3 and 4 are considered normal and ideal for digestive health.
Time to oral nutrition | Measured up to 90 days from randomization
  This is defined as the cessation of tube feeding and it serves as an important metric in evaluating patients with EPI, as it may act as a surrogate measure for the restoration of adequate digestive function.

CONTACTS AND LOCATIONS:
Overall Officials: Casey M Luckhurst, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stevens J, Wyatt C, Brown P, Patel D, Grujic D, Freedman SD. Absorption and Safety With Sustained Use of RELiZORB Evaluation (ASSURE) Study in Patients With Cystic Fibrosis Receiving Enteral Feeding. J Pediatr Gastroenterol Nutr. 2018 Oct;67(4):527-532. doi: 10.1097/MPG.0000000000002110. PMID 30074573
- [Background] Johnson CD, Williamson N, Janssen-van Solingen G, Arbuckle R, Johnson C, Simpson S, Staab D, Dominguez-Munoz E, Levy P, Connett G, Lerch MM. Psychometric evaluation of a patient-reported outcome measure in pancreatic exocrine insufficiency (PEI). Pancreatology. 2019 Jan;19(1):182-190. doi: 10.1016/j.pan.2018.11.013. Epub 2018 Nov 27. PMID 30528109
- [Background] Johnson CD, Arbuckle R, Bonner N, Connett G, Dominguez-Munoz E, Levy P, Staab D, Williamson N, Lerch MM. Qualitative Assessment of the Symptoms and Impact of Pancreatic Exocrine Insufficiency (PEI) to Inform the Development of a Patient-Reported Outcome (PRO) Instrument. Patient. 2017 Oct;10(5):615-628. doi: 10.1007/s40271-017-0233-0. PMID 28332032